CLINICAL TRIAL: NCT02223728
Title: Evaluation of Telehealth Lifestyle Program for Persons With Traumatic Brain Injury: Objective 2
Brief Title: Evaluation of a Telehealth Lifestyle Management Program to Improve Healthy Behaviors Post Head Injury
Acronym: ProjectLIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laura E. Dreer, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H133A120096; H133A120096 (Other Grant/Funding Number: H133A120096)
Record Dates: First submitted 2014-08-19; First posted 2014-08-22 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Condition (Experimental): Telehealth Lifestyle Program
  Interventions: Behavioral: Lifestyle
- Attention Control Condition (Sham Comparator): Health Education Program
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Lifestyle
  Arms: Treatment Condition
Behavioral: Health Education
  Arms: Attention Control Condition

SUMMARY:
Interventions to help individuals with traumatic brain injury manage their healthy lifestyle behaviors have been limited. Thus, the goal of this project is to evaluate the efficacy of a telehealth lifestyle program on reductions in weight and improvements in health behaviors/lifestyle choices.

ELIGIBILITY:
Inclusion Criteria:

1. age 19 years or older
2. English speaking
3. sustained a moderate or severe TBI (as defined by a period of confusion after the injury of more than 24 hours)
4. overweight or obese as defined by a BMI score of ≥ 25 kg/m2
5. 1-year or greater post-injury
6. not currently enrolled in a weight loss program or receiving weight loss medication
7. regular access to a computer/laptop with internet capability which allows internet and telephone access simultaneously
8. if person with TBI who meets criteria 1-7 but does not cook, shop, and/or prepare meals independently, he or she must have a non-paid, study partner willing to participate in the study.

Exclusion Criteria:1

1. pregnant or planning to become pregnant in the next 7 months
2. concurrent medical condition for which changes in exercise or diet would be contraindicated
3. severe hearing or visual impairment
4. significant psychiatric disorder, such as schizophrenia or bipolar disorder (those with depression or anxiety will not be excluded)
5. unable to communicate
6. significant cognitive impairment and without a study partner, and/or
7. person with TBI who does not cook, shop, and/or prepare meals independently who does not have a non-paid, study partner willing to participate in the study
8. currently enrolled in an organized weight loss program
9. has lost > 10% of body weight over the past 6 months
10. history of an eating disorder

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-08; Primary Completion 2018-10 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) scores | Changes in baseline and post-program BMI scores at 7-months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dreer, Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham/Spain Rehabilitation Center, Birmingham, Alabama, United States